CLINICAL TRIAL: NCT06282354
Title: Telemedicine for Postoperative Follow-up After Oncological Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: NP4035/2023
Record Dates: First submitted 2024-01-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Urologic Cancer; Satisfaction, Patient; Surgery; Postoperative Adhesion
MeSH Terms: conditions — Urologic Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Face-to-face appointment: Patients allocated in face-to-face appointment after urooncologic surgical procedures
  Interventions: Other: Type of post-operative appointment
- Telemedicine appointment: Patients allocated in telemedicine appointment after urooncologic surgical procedures
  Interventions: Other: Type of post-operative appointment

INTERVENTIONS:
Other: Type of post-operative appointment — remote post-operative appointment for small or medium urooncology procedures

SUMMARY:
The study will be a prospective, randomized, non-inferiority, open-label study, to be carried out at the Cancer Institute of the State of São Paulo for 6 months and will include patients agreeing to voluntary participation upon signing an informed consent form.

DETAILED DESCRIPTION:
All patients with urological neoplasms who have undergone low and medium complexity surgical procedures (e.g. prostate TUR, Bladder TURP, double-J passage, partial or total videolaparoscopic and open nephrectomies) at ICESP will be invited to participate. It will be excluded all patients undergoing emergency operations, outpatient procedures, major procedures, patients with probes or drains or no support for home telemedicine.A telemedicine platform for video conferencing will be used by the healthcare team at our institution. The information from the patient will be protected by security passwords following ethical and legal provisions.

The patient will be invited to participate in the study at the preoperative evaluation. If it agrees to participate, it will sign the agreement informed consent, and will be randomized in the Redcap® software to one of the study arms (post-operative consultations in person or telemedicine). Patient follow-up in the study will be carried out with the first post-surgery visit between 10 - 20 days after discharge, according to the type of consultation for which the patient was randomized pre-surgery. The main outcome assessed will be the degree of patient satisfaction assessed by using a Likert scale. For patients randomized to the telemedicine arm, the global perception of satisfaction in all aspects of the teleconsultation will be quantified through a Patient Satisfaction Assessment questionnaire served via telemedicine. It will also be evaluated the perception of security defined as security of personal information (Laws General Data Protection - LGPD) . For patients randomized to the in-person postoperative consultations arm, it will be applied an adapted questionnaire, based on QAS-Tele, in order to verify the degree of patient satisfaction in relation to their type of consultation and their interest in carrying out telemedicine consultations in the future.

Questionnaires will be administered to patients 5 to 10 days after the first post-operative return to evaluate the issues mentioned by members of the research team via telephone contact. In addition to this information, patients coming to the institution's emergency room will be quantified within a period of up to 30 days after surgery.

The secondary outcomes will be the number of unattended arrivals programmed at the institution, presence of postoperative complications graded according to the Clavien-Dindo classification, appointment's duration, number of exams requested by the attending physicians, total cost involved per service (expenses with travel, mobile internet data package, necessary structure to telemedicine services) and environmental impact generated with both types of services. Patients will have their demographic data and clinical conditions recorded in appropriate database using RedCap software (Sex, Age, index of body mass, classification of the American Society of Anesthesiologists, Charlson classification, Clavien-Dindo classification). The descriptive analysis will be made by reporting the quantitative variables through the mean, standard deviation, median and quartile, and statistical analysis performed using the Wilcoxon-Mann-Whitney.

ELIGIBILITY:
Inclusion Criteria:

* All patients with urological neoplasms who have undergone low and medium complexity surgical procedures (e.g. prostate TUR, Bladder TURP, double-J passage, partial or total nephrectomy videolaparoscopic and open) at ICESP

Exclusion Criteria:

* All patients undergoing emergency operations, outpatient procedures, major procedures, patients with probes or drains or no support for home telemedicine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Oncologic patients from the ICESP
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction in the post-operative return | 10 - 20 days after the surgical procedure
  Degree of patient satisfaction assessed by using a Likert scale with seven questions about the appointment quality and grading with five answers (definitely not, probably not, maybe, probably yes, definitely yes)

SECONDARY OUTCOMES:
unattended arrivals at the institution | 30 days
  Number of unattended arrivals at the institution or emergency services
Postoperative complications | 30 days
  Presence of postoperative complications graded according to the Clavien-Dindo classification
Appointment's time | 30 days
  Duration of the appointment
Number of exams requested | 10 - 20 days
  Number of exams requested by the attending physicians in the post-operative return
Total cost involved per service | 10 - 20 days
  Expenses with travel, mobile internet data package, necessary structure to telemedicine services
Environmental impact | 10 - 20 days
  Environmental impact in the follow-up measured by carbon dioxide emission produced by the type of transportation and travel time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heymann DL, Shindo N; WHO Scientific and Technical Advisory Group for Infectious Hazards. COVID-19: what is next for public health? Lancet. 2020 Feb 22;395(10224):542-545. doi: 10.1016/S0140-6736(20)30374-3. Epub 2020 Feb 13. No abstract available. PMID 32061313
- [Background] Lerner AM, Folkers GK, Fauci AS. Preventing the Spread of SARS-CoV-2 With Masks and Other "Low-tech" Interventions. JAMA. 2020 Nov 17;324(19):1935-1936. doi: 10.1001/jama.2020.21946. No abstract available. PMID 33104157
- [Background] Walker J, Fleece ME, Griffin RL, Leal SM, Alsip JA, Stigler WS, Nafziger SD, Marrazzo JM, Lee RA. Decreasing High-risk Exposures for Healthcare Workers Through Universal Masking and Universal Severe Acute Respiratory Syndrome Coronavirus 2 Testing on Entry to a Tertiary Care Facility. Clin Infect Dis. 2021 Nov 2;73(9):e3113-e3115. doi: 10.1093/cid/ciaa1358. PMID 32901247
- [Background] Loeb AE, Rao SS, Ficke JR, Morris CD, Riley LH 3rd, Levin AS. Departmental Experience and Lessons Learned With Accelerated Introduction of Telemedicine During the COVID-19 Crisis. J Am Acad Orthop Surg. 2020 Jun 1;28(11):e469-e476. doi: 10.5435/JAAOS-D-20-00380. PMID 32301818
- [Background] Ohannessian R, Duong TA, Odone A. Global Telemedicine Implementation and Integration Within Health Systems to Fight the COVID-19 Pandemic: A Call to Action. JMIR Public Health Surveill. 2020 Apr 2;6(2):e18810. doi: 10.2196/18810. PMID 32238336
- [Background] Committee on Improving the Quality of Cancer Care: Addressing the Challenges of an Aging Population; Board on Health Care Services; Institute of Medicine; Levit L, Balogh E, Nass S, Ganz PA, editors. Delivering High-Quality Cancer Care: Charting a New Course for a System in Crisis. Washington (DC): National Academies Press (US); 2013 Dec 27. Available from http://www.ncbi.nlm.nih.gov/books/NBK202148/ PMID 24872984
- [Background] Kummerow Broman K, Roumie CL, Stewart MK, Castellanos JA, Tarpley JL, Dittus RS, Pierce RA. Implementation of a Telephone Postoperative Clinic in an Integrated Health System. J Am Coll Surg. 2016 Oct;223(4):644-51. doi: 10.1016/j.jamcollsurg.2016.07.010. Epub 2016 Aug 18. PMID 27545100
- [Background] Nikolian VC, Williams AM, Jacobs BN, Kemp MT, Wilson JK, Mulholland MW, Alam HB. Pilot Study to Evaluate the Safety, Feasibility, and Financial Implications of a Postoperative Telemedicine Program. Ann Surg. 2018 Oct;268(4):700-707. doi: 10.1097/SLA.0000000000002931. PMID 30095477
- [Background] Moreira TC, Constant HM, Faria AG, Matzenbacher AMF, Balardin GU, Matturro L, Silva MS, Umpierre RN, Rodrigues AS, Cabral FC, Pagano CGM. Tradução, adaptação transcultural e validação de questionário de satisfação em telemedicina. Rev Bras Med Fam Comunidade. 2022;17(44):2837.